CLINICAL TRIAL: NCT03163056
Title: Behavioral Activation and Voucher-based Contingency Management for Smokers With Depression
Brief Title: Smoking Cessation Treatment for Depressed Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Roberto Secades, Professor/PhD, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSI2015-64371-P
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking cessation; Depression; Clinical trial
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to each of the three treatment conditions in accordance with a computer-generated randomization list. The three treatment conditions will be actively running in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-behavioral treatment (CBT) (Other): The CBT treatment condition is implemented in group-based sessions carried out during 8 weeks. Components included: information about tobacco, behavioral contract whereby patients committed to attend sessions, self-monitoring and graphical representation of cigarette smoking, nicotine fading (a weekly reduction of 30% of nicotine intake from the first to the four week, and abstinence from the fifth week onwards), physiological feedback (CO in expired air and cotinine analyses) on cigarette intake, stimulus control, strategies for managing nicotine withdrawal symptoms, training in alternative behaviors, and relapse prevention strategies (e.g., problem solving techniques).
  Interventions: Behavioral: Cognitive-behavioral treatment (CBT)
- CBT+Behavioral Activation (BA) (Active Comparator): This intervention includes both CBT and BA strategies for smoking cessation and depression management. Participants allocated to this condition received 8 therapy sessions. The BA module included: treatment rationale, information on the relationship between smoking and depression, identification of life areas, values and activities, generation of meaningful and reinforcing activities, social support (i.e., behavioral contracts).
  Interventions: Behavioral: Cognitive-behavioral treatment (CBT); Behavioral: CBT+Behavioral Activation (BA)
- CBT+BA+ Contingency Management (CM) (Active Comparator): This intervention is provided in the same manner as the above treatment protocols but with the addition of a CM procedure reinforcing abstinence since fifth session and onwards. The number of sessions was the same as in the aforementioned treatment conditions and CO and cotinine samples were also collected. Participants providing negative specimens of both CO (≤4 ppm) and cotinine (≤80 ng/ml) earned points exchangeable for rewards (e.g., cinema tickets) on a schedule of escalating magnitude of reinforcement (from 10€ voucher value with maximum possible earnings of 175€ in vouchers).
  Interventions: Behavioral: Cognitive-behavioral treatment (CBT); Behavioral: CBT+Behavioral Activation (BA); Behavioral: CBT+BA+ Contingency Management (CM)

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment (CBT) — The CBT was implemented in group-based sessions of four patients. Sessions were carried out once a week over a 8-week period, with quite date occurring at fifth session. The main component was nicotine fading. From the first to the fourth week, patients were asked to gradually reduce their nicotine intake based on a weekly reduction of 30%. A maximum number of cigarettes per day and also specific cigarette brands with lower nicotine levels were recommended. Other components of the CBT program included information about tobacco, a behavioral contract, self monitoring and graphical representation of cigarette smoking, stimulus control, strategies for controlling nicotine withdrawal symptoms, physiological feedback, training in alternative behaviors, and relapse prevention strategies.
Behavioral: CBT+Behavioral Activation (BA) — This intervention was provided as in the above CBT condition, that is, eight group-based sessions of four patients. Nevertheless, this treatment included a BA component for addressing both smoking cessation and depression management. The BA module included: treatment rationale, information on the relationship between smoking and depression, identification of life areas, values and activities, generation of meaningful and reinforcing activities, social support (i.e., behavioral contracts).
  Arms: CBT+BA+ Contingency Management (CM); CBT+Behavioral Activation (BA)
Behavioral: CBT+BA+ Contingency Management (CM) — This intervention was provided in the same manner as the above mentioned treatment protocols but with the addition of a contingency management procedure reinforcing abstinence since fifth session and onwards. The number of sessions was the same as in the aforementioned treatment conditions and CO and cotinine samples were also collected. Participants providing negative specimens of both CO (≤4 ppm) and cotinine (≤80 ng/ml) earned points exchangeable for rewards (e.g., cinema tickets) on a schedule of escalating magnitude of reinforcement (from 10€ voucher value with maximum possible earnings of 175€ in vouchers).
  Arms: CBT+BA+ Contingency Management (CM)

SUMMARY:
The present research project aims to develop an innovative and empirically validated intervention protocol for smoking cessation among patients with depressive symptoms. For this purpose, two smoking cessation treatments tailored for managing depression will be compared with a standard smoking cessation treatment. Participants will be assigned to one of the following three treatment conditions: 1) Cognitive-behavioral treatment for smoking cessation (CBT); 2) CBT plus Behavioral Activation (BA); 3) CBT+BA+ Contingency Management (CM).

The main goals are:

1. To assess abstinence rates in each of the above-mentioned treatment conditions conditions at short and long-term follow-ups: post-treatment, once during the first three months, and at at six after post-treatment.

1. To assess the effectiveness (relapse rate) of each treatment condition at short and long-term follow-ups: post-treatment, once during the first three months,and at six after post-treatment.

3. To analyze efficiency (cost-efficacy) and feasibility of the treatments to a community setting.

4. To analyze the moderating effect of individual variables over treatment outcomes. In particular, moderating variables will be: sociodemographic characteristics, severity of nicotine dependence, severity of depressive symptomatology and impulsivity.

The study hypothesis are:

1-Adding a voucher-based CM component to CBT+BA will enhance abstinence rates and decrease both short and long-term relapse rates.

2. Providing smoking cessation treatments that include a mood management component (BA or BA+CM) will have a positive impact in ameliorating depression.

3. Certain individual variables (e.g., gender, nicotine dependence and depression severity and impulsivity) will have a moderating effect on treatment outcomes.

4. Both CBT+BA and CBT+BA+CM will prove cost-effectiveness and thus may be generalized to a clinical and community context.

DETAILED DESCRIPTION:
Cigarette smoking continues to have a startling adverse impact on public health, leading to more than 5 million premature deaths annually worldwide. Smoking rates are disproportionately high among the population suffering from depression. In this regard, smokers with comorbid depression are more likely to smoke heavily and meet criteria for high nicotine dependence. It is also more probable that they experience negative mood changes after withdrawal and show shorter time to relapse and lower rates of abstinence when attempting to quit compared to non-depressed smokers. In recent years there has been a great interest in developing effective strategies to promote abstinence in smokers with depression. In particular, a proliferation on Behavioral Activation (BA) treatments for smokers with depression has been recently produced. There is promising evidence for the positive effect of BA treatments upon both quitting smoking and depression. On the other hand, Contingency Management (CM) has shown promising results in promoting both retention and nicotine abstinence among comorbid and non-comorbid smokers. Nevertheless, there is a lack of research exploring the effectiveness of CM on smokers with depression.

The primary aim of this clinical trial is to yield data on the effectiveness of BA and CM for smoking cessation in smokers with depression. To address this issue, both BA and CM interventions will be compared with a standard smoking cessation treatment, namely Cognitive-behavioral treatment (CBT) for smoking cessation. Participants will be assigned to one of the following three treatment conditions: 1) Cognitive-behavioral treatment for smoking cessation (CBT); 2) CBT plus Behavioral Activation (BA); 3) CBT+BA+Contingency Management (CM).

Regarding the factors contributing to improve the quality of the present clinical trial, sample size was estimated using the software G*Power 3.1. An estimated sample size of 150 participants would detect a medium effect size (Cohen's d = 0.3, with power (1-β) set at 0.97 and α = 05).

Given that data will be collected up to six months after post-treatment, moderate rates of lost to follow-up can be expected. However, the sample size estimate in this study will be sufficient to ensure a representative distribution of the population to whom results will be generalized.

The primary analyses derived from this clinical trial will be conducted using Statistical Package for the Social Science (SPSS) version 22 for Windows. A set of descriptive and frequency analyses will be carried out with regard to the participants' characteristics. Comparisons between the treatment groups for baseline characteristics will be conducted using t-tests for independent groups. A set of chi-square tests for categorical variables, and independent samples t-tests (two-tailed) for continuous variables (after Levene's correction for inequality of variance) will be performed to examine the main effect of each treatment condition on abstinence and relapse rates.

ELIGIBILITY:
Inclusion Criteria:

* being age 18 or over
* having smoked 10 or more cigarettes/day within the last year
* meeting criteria for current unipolar major depression disorder according to the Diagnostic and Statistical Manual of Mental Disorders-4th ed., text rev (DSM-IV-TR) (American Psychiatric Association 2000).

  , and/or scoring ≥ 14 on the Beck Depression Inventory (Beck, Steer, & Brown, 1996)
* meeting the diagnostic criteria for nicotine dependence according to the Diagnostic and Statistical Manual of Mental Disorders-4th ed., text rev (DSM-IV-TR) (American Psychiatric Association 2000).

Exclusion Criteria:

* not being able to attend the entire treatment,
* suffering from severe mental disorders others than depression such as cognitive impairment, a psychotic disorder or bipolar disorder.
* being currently receiving other psychological treatment for smoking cessation or depression.
* meeting criteria for abuse and/or dependence on a substance other than nicotine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | end of treatment (8-week)
  Abstinence is considered when participants met the following criterion: 24-hours point prevalence abstinence. Abstinence is confirmed by asking participants to provide a sample of carbon monoxide (CO) and cotinine urine.
smoking abstinence | 1 month follow-up
  Abstinence is considered when participants met the following criterion: 7-day point prevalence abstinence. Abstinence is confirmed by asking participants to provide a sample of carbon monoxide (CO) and cotinine urine.
smoking abstinence | 2 months follow-up
  Abstinence is considered when participants met the following criterion: 7-day point prevalence abstinence. Abstinence is confirmed by asking participants to provide a sample of carbon monoxide (CO) and cotinine urine.
smoking abstinence | 3 months follow-up
  Abstinence is considered when participants met the following criterion: 7-day point prevalence abstinence. Abstinence is confirmed by asking participants to provide a sample of carbon monoxide (CO) and cotinine urine.
smoking abstinence | 6 months follow-up
  Abstinence is considered when participants met the following criterion: 7-day point prevalence abstinence. Abstinence is confirmed by asking participants to provide a sample of carbon monoxide (CO) and cotinine urine.

SECONDARY OUTCOMES:
depression | intake (baseline), end of treatment (8-week),1,2,3 and 6 months follow-up
  Changes in depression are assessed using the Beck's Depression Inventory- Second Edition (BDI-II). Scores are examined as a continuous scale. None/minimal depression is defined as scoring below the clinical screening BDI cutoff of mild depression (<14). Depression diagnosis is assessed in those individuals scoring 14 or more on the BDI-II by means of the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders-Clinical Version (SCID-I/CV).
behavioral activation | intake (baseline), end of treatment (8-week),1,2,3 and 6 months follow-up
  In order to assess behavioral activation, we use the Behavioral Activation for Depression Scale-Short Form (BADS-SF) (Kanter, Mulick, Busch, & Martell, 2012). This instrument can be used to track changes weekly in the behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation. It examines changes in the following areas: activation, avoidance/rumination, work/school impairment, and social impairment. The BADS-SF consists of 9 questions, each rated on a seven point scale ranging from 0 (not at all) to 6 (completely).
environmental reward | intake (baseline), end of treatment (8-week),1,2,3 and 6 months follow-up
  The Environmental Reward Observation Scale (EROS)(Barraca & Pérez-Álvarez, 2010) is used to assess this outcome.The EROS is a brief, reliable and valid measure of environmental reward that improves the psychological assessment of negative mood states such as clinical depression. It consists of 10 items rated on a four point scale ranging from 1 (completely disagree) to 4 (completely agree).
cigarette craving | intake (baseline), end of treatment (8-week),1,2,3 and 6 months follow-up
  The Questionnaire of smoking urges (QSU-Brief) (Cox, Tiffany & Christen, 2001) is used to assess cigarette craving. This 10-item, self-report instrument provides an adequate assessment of multiple aspects of cigarette craving. All items are rated on a seven point scale raging from 1 (completely disagree) to 7 (completely agree). Factor analyses revealed that this instrument has a two-factor solution. The first factor reflects a strong desire and intention to smoke, with smoking perceived as rewarding for active smokers. The second factor represents an anticipation of relief from negative affect with an urgent desire to smoke.
anxiety | intake (baseline), end of treatment (8-week),1,2,3 and 6 months follow-up
  To assess anxiety levels, we use the State-Trait Anxiety Inventory (STAI) (Spielberger, Gorsuch, Lushene, Vagg & Jacobs, 1983). This is a widely used self-report instrument that assesses the presence and severity of current symptoms of anxiety and a generalized propensity to be anxious. There are two subscales within this measure. The first is the the State Anxiety Scale (S-Anxiety) that evaluates the current state of anxiety. The second is the Trait Anxiety Scale (T-Anxiety) that evaluates relatively stable aspects of "anxiety proneness," including general states of calmness, confidence, and security. It has 40 items, 20 items allocated to each of the S-Anxiety and T-Anxiety subscales. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always").
impulsivity | intake (baseline), end of treatment (8-week),1,2,3 and 6 months follow-up
  Impulsivity levels are assessed by means of the delay discounting task. Participants complete a computerized version of this task. They are presented with several choices, ranging from notionally being given €1,000 after a fixed delay, versus various amounts of money given immediately using an adjusting-amount procedure (Holt, Green, & Myerson, 2012). The delay values used are one day, one week, one month, six months, one year, five years, and 25 years. Delay discounting is calculated using logk and the area under the curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Secades-Villa, PhD, Principal Investigator — University of Oviedo
Locations (1):
- Clinical Unit of Addictive Behaviors, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Secades-Villa R, Garcia-Rodriguez O, Lopez-Nunez C, Alonso-Perez F, Fernandez-Hermida JR. Contingency management for smoking cessation among treatment-seeking patients in a community setting. Drug Alcohol Depend. 2014 Jul 1;140:63-8. doi: 10.1016/j.drugalcdep.2014.03.030. Epub 2014 Apr 8. PMID 24768410
- [Background] MacPherson L, Tull MT, Matusiewicz AK, Rodman S, Strong DR, Kahler CW, Hopko DR, Zvolensky MJ, Brown RA, Lejuez CW. Randomized controlled trial of behavioral activation smoking cessation treatment for smokers with elevated depressive symptoms. J Consult Clin Psychol. 2010 Feb;78(1):55-61. doi: 10.1037/a0017939. PMID 20099950
- [Background] van der Meer RM, Willemsen MC, Smit F, Cuijpers P. Smoking cessation interventions for smokers with current or past depression. Cochrane Database Syst Rev. 2013 Aug 21;(8):CD006102. doi: 10.1002/14651858.CD006102.pub2. PMID 23963776
- [Background] Secades-Villa R, Vallejo-Seco G, Garcia-Rodriguez O, Lopez-Nunez C, Weidberg S, Gonzalez-Roz A. Contingency management for cigarette smokers with depressive symptoms. Exp Clin Psychopharmacol. 2015 Oct;23(5):351-60. doi: 10.1037/pha0000044. Epub 2015 Aug 17. PMID 26280589
- [Derived] Notley C, Gentry S, Livingstone-Banks J, Bauld L, Perera R, Conde M, Hartmann-Boyce J. Incentives for smoking cessation. Cochrane Database Syst Rev. 2025 Jan 13;1(1):CD004307. doi: 10.1002/14651858.CD004307.pub7. PMID 39799985
- [Derived] Gonzalez-Roz A, Weidberg S, Garcia-Perez A, Martinez-Loredo V, Secades-Villa R. One-Year Efficacy and Incremental Cost-effectiveness of Contingency Management for Cigarette Smokers With Depression. Nicotine Tob Res. 2021 Jan 22;23(2):320-326. doi: 10.1093/ntr/ntaa146. PMID 32772097
- [Derived] Weidberg S, Secades-Villa R, Garcia-Perez A, Gonzalez-Roz A, Fernandez-Hermida JR. The synergistic effect of cigarette demand and delay discounting on nicotine dependence among treatment-seeking smokers. Exp Clin Psychopharmacol. 2019 Apr;27(2):146-152. doi: 10.1037/pha0000248. Epub 2018 Dec 20. PMID 30570273